CLINICAL TRIAL: NCT00359541
Title: Voriconazole Plasma Concentration and Toxicity
Brief Title: Voriconazole Blood Levels and Toxicity
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060077; 06-I-0077
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-06-25

CONDITIONS: Pharmacology
Keywords: CYP2C9; CYP2C19; Pharmacology; Genotype; Metabolism

SUMMARY:
This study will look at how voriconazole, a drug used to treat or protect against fungal infections, affects the body. Adverse effects associated with voriconazole include skin problems and temporary changes in vision, mental status and liver function. There is some evidence that these side effects may be more intense when there are high levels of the drug in the blood. The amount of voriconazole in the body is determined by how much of the drug the patient receives and by the patient's ability to inactivate and excrete it, which may be determined in part by genes. This study will examine: 1) side effects patients develop from voriconazole; 2) whether the side effects experienced are related to the concentration of drug in the body; and 3) the role of genes in determining how quickly the body inactivates and excretes the drug.

Patients 12 and older who are participating in studies in the National Institute of Allergy and Infectious Diseases (NIAID), the National Cancer Institute (NCI) or the National Heart, Lung, and Blood Institute (NHLBI) and have been treated with voriconazole for 15 days or less may be eligible for this study.

Participation involves the following:

* Identification and recording of adverse effects patients experience due to voriconazole treatment
* Collection of basic information about the patient's medical history and treatment
* Blood draws once a week during the patient's hospitalization
* Collection of routine laboratory test results ordered by the patient's doctor
* Blood draw to identify genes responsible for voriconazole inactivation
* Weekly monitoring for the possibility of voriconazole adverse effects
* Blood draw to measure blood levels of voriconazole when the drug is stopped, if it is stopped because of an adverse effect
* Evaluations at outpatient visits, including a blood draw to measure voriconazole blood levels

Participation in the study ends 7 days after voriconazole treatment is stopped because it is no longer needed.

DETAILED DESCRIPTION:
Voriconazole (Vfend(Registered Trademark), Pfizer) has achieved common usage at the NIH (National Institutes of Health) Clinical Research Center for the treatment of fungal infections in immunosuppressed patients. Toxicity includes relatively frequent but reversible changes in vision and more infrequent, potentially serious hepatotoxicity, decreased cognitive function and rash. Incidence of these more serious adverse events has been difficult to ascertain because of the morbidity of underlying disease in patients receiving voriconazole, but a minimum estimate is 10 percent. It is known that voriconazole plasma concentrations vary between patients over a fifty-fold range but it is not known whether toxicity is related to plasma drug exposure. The reason for the differing voriconazole plasma concentrations between normal individuals is partly due to genetic variations in hepatic cytochrome enzymes CYP2C9 and CYP2C19 (Cytochrome P450, family 2, subfamily C, polypeptide 9 and 19, respectively). In patients with underlying illness, drug interactions and decreased hepatic drug clearance may contribute to variability.

The purpose of the study is to record prospectively the adverse effects of voriconazole in Clinical Center patients who have been prescribed the drug by their primary physician. We will ask the primary physician to order a trough voriconazole plasma levels once a week. The test will not be reported to the physician. Because interpretation of the test is unknown, the physicians will be blinded to the report. Rather, the primary objective of the study is to analyze the voriconazole plasma concentrations when the study is completed to determine if there is a concentration and duration of drug exposure that correlates with toxicity. A secondary objective is to determine the 2C9 and 2C19 genotype of patients and search for possible correlations between genotype and plasma voriconazole concentrations. Administration of other drugs given to the patient will be tracked to analyze whether any previously unknown drug interactions seem to have changed the voriconazole plasma concentration. The study will also determine the incidence of adverse effects of voriconazole in our patient population.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients, at least 12 years old with no restriction of gender, race or disabilities, followed by the National Institute of Allergy and Infectious Diseases (NIAID), National Cancer Institute (NCI) and National Heart Lung and Blood Institute (NHLBI) who begin treatment with voriconazole either oral or intravenous.

Patients who have a previous voriconazole course at least 7 days before current course.

EXCLUSION CRITERIA:

Time elapsed greater than 15 days from initiation of voriconazole treatment for inpatients and greater than 30 days from initiation of voriconazole treatment for outpatients.

Patients who the medical staffs caring for the patient not want entered into the study.

Patients unable to give informed consent, due to the severity of their medical condition (Comatose patients, ICU patients under sedation).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-01-19; Study Completion 2010-06-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jantunen E, Ruutu P, Niskanen L, Volin L, Parkkali T, Koukila-Kahkola P, Ruutu T. Incidence and risk factors for invasive fungal infections in allogeneic BMT recipients. Bone Marrow Transplant. 1997 Apr;19(8):801-8. doi: 10.1038/sj.bmt.1700737. PMID 9134172
- [Background] Herbrecht R, Denning DW, Patterson TF, Bennett JE, Greene RE, Oestmann JW, Kern WV, Marr KA, Ribaud P, Lortholary O, Sylvester R, Rubin RH, Wingard JR, Stark P, Durand C, Caillot D, Thiel E, Chandrasekar PH, Hodges MR, Schlamm HT, Troke PF, de Pauw B; Invasive Fungal Infections Group of the European Organisation for Research and Treatment of Cancer and the Global Aspergillus Study Group. Voriconazole versus amphotericin B for primary therapy of invasive aspergillosis. N Engl J Med. 2002 Aug 8;347(6):408-15. doi: 10.1056/NEJMoa020191. PMID 12167683
- [Background] Walsh TJ, Pappas P, Winston DJ, Lazarus HM, Petersen F, Raffalli J, Yanovich S, Stiff P, Greenberg R, Donowitz G, Schuster M, Reboli A, Wingard J, Arndt C, Reinhardt J, Hadley S, Finberg R, Laverdiere M, Perfect J, Garber G, Fioritoni G, Anaissie E, Lee J; National Institute of Allergy and Infectious Diseases Mycoses Study Group. Voriconazole compared with liposomal amphotericin B for empirical antifungal therapy in patients with neutropenia and persistent fever. N Engl J Med. 2002 Jan 24;346(4):225-34. doi: 10.1056/NEJM200201243460403. PMID 11807146